CLINICAL TRIAL: NCT07118202
Title: TheraBionic P1 Device for Patients With Advanced Hepatocellular Carcinoma (HCC) Who Fail First and Second Line Therapy
Brief Title: TheraBionic P1 Device in Subjects With Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: THERABIONIC INC. (Other)
Responsible Party: Principal Investigator, Anthony F. Shields, MD PhD, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-074
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma Recurrent

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TheraBionic P1 device (Experimental): Self administered Amplitude-modulated electromagnetic fields three times daily
  Interventions: Device: TheraBionic P1

INTERVENTIONS:
Device: TheraBionic P1 — Amplitude-modulated electromagnetic fields will be self-administered and given continuously to patients in three 60-minute treatments per day, administered in the morning, middle of the day, and in the evening

SUMMARY:
The goal of this clinical trial is to learn if the TheraBionic P1 device given to patients with advanced hepatocellular carcinoma (HCC) who have no standard of care options can affect patients survival. The main questions it aims to answer are:

* will the TheraBionic P1 device affect overall survival in advance HCC
* the long term safety and tolerability of the TheraBionic P1 device
* assessment of how the disease responded to the TheraBionic P1 device

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced hepatocellular carcinoma (HCC) (defined as a liver tumor not eligible for local therapies given the extent of disease or a livor tumor that recurred after local therapy)
* Patients who have failed at least two lines of therapy* or who are no longer eligible for any line of standard therapy or who are intolerant to at least two lines of therapy.
* Patients with pacemakers or other implantable devices may be treated with the TheraBionic P1 device.
* Patients must be ≥ 22 years old and must be able to understand and sign an informed consent.
* Female patients of childbearing potential and their partners and male patients must agree to use adequate contraception during the period of study treatment.
* Patients with a life expectancy of at least 3 months

Exclusion Criteria:

* Oral mucosa is not intact (i.e., case of mucositis, thrush, bleeding mucosal lesions, oral herpes, aphthous stomatitis, mouth ulcers, canker sores or gingivostomatitis, herpangina, aphthae).
* Patients receiving calcium channel blockers and any agent blocking L-type of T-type Voltage Gated Calcium Channels, e.g., amlodipine, nifedipine, ethosuximide, ascorbic acid (vitamin C), etc. unless their medical treatment is modified to prior to enrollment exclude calcium channel blockers for the duration of treatment on study. (Refer to Appendix B for a comprehensive list of excluded medications)
* Patients that do not agree to be followed according to the study protocol or have cognitive or physical inability to use the device.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From start of treatment until death, up to 24 months
  Overall survival assessment will be recorded in days and will represent the period starting at the date of treatment initiation and finishing at the date of patient death from any cause.
  Living patients at the time of analysis will have the date of last contact (consultation visit or phone contact) used to define overall survival

SECONDARY OUTCOMES:
PROMIS Measures of Pain Interference | From Start of Treatment to the end of treatment up to 12 months
  National Institutes of Health Patient Reported Outcome Measurement Information System (PROMIS) measures of Pain Interference short form 4a. PROMIS scores can range from 0 to 100; scales are calibrated using a T-score metric with a mean of 50 and standard deviation of 10. A higher score indicates more pain interference (poorer health). 4 items
Patient-reported outcomes (PRO) | From Start of Treatment to the end of treatment up to 12 months
  Patient-reported outcomes (PRO) measures will assess the trajectory of patient rated tolerability of treatment (Functional Assessment of Cancer Therapy items regarding bother of side effects, one item), patient-rated symptomatic adverse events (11 Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events item library items)
PROMIS Measures of Pain Intensity | From Start of Treatment to the end of treatment up to 12 months
  NIH Patient Reported Outcome Measurement Information System (PROMIS) measures of Pain Intensity short form 1a. PROMIS scores can range from 0 to 100; scales are calibrated using a T-score metric with a mean of 50 and standard deviation of 10. A higher score indicates more pain intensity (poorer health). 1 item
ECOG Performance Status | From Start of Treatment to the end of treatment up to 12 months
  (ECOG)Eastern Cooperative Oncology Group performance status scale to measure functional status and ability to carry out activities of daily living. A system used to assess how a patient's cancer or other serious illness affects their daily living abilities. It's a 6-point scale (0-5) where lower scores indicate better function and higher scores indicate more limitations
Disease Control Rate | From enrollment up to 6 months
  Disease control will be defined as the percentage of patients who are alive and have documented response status of complete response (CR), partial response (PR) or stable disease (SD) at 4 months and 6 months from the date of enrollment.
Duration of overall response | From start of treatment up to 24 months
  Measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded on study).
  The duration of overall complete response is measured from the time measurement criteria are first met for CR until the first date that recurrent disease is objectively documented. Duration of stable disease: Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started
Time to Progression (TTP) | Start of treatment to death from any cause up to 24 months
  Time-to-radiological progression assessment will be recorded in days and will represent the period starting at the date of treatment initiation and finishing at the date of radiological assessment documenting tumor progression. Patients who initiate post-study anticancer therapy or die without documented progression will be censored at that time point.
Progression-free survival (PFS) | Start of treatment to progression of disease, last follow-up on study or death, whichever comes first up to 24 months
  Progression-free survival assessment will be recorded in days and will represent the period starting at the date of treatment initiation and finishing at the later of the date of documentation of radiologic tumor progression, date of last follow-up on study treatment or death, whichever comes first. Patients who initiate post-study antitumor therapy prior to radiologic progression will be censored for PFS at that date.
PROMIS Measures of Physical Function | From Start of Treatment to the end of treatment up to 12 months
  National Institutes of Health Patient Reported Outcome Measurement Information System (PROMIS) measures of physical function short form 4a. PROMIS scores can range from 0 to 100; scales are calibrated using a T-score metric with a mean of 50 and standard deviation of 10. A higher score indicates less physical function (poorer health). 4 items

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F Shields, M.D., Principal Investigator — Wayne State University
Locations (6):
- United States (6):
  - Karmanos Cancer Institute at McLaren Bay Region, Bay City, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute at McLaren Flint, Flint, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Karmanos Cancer Institute at McLaren Lapeer Region, Lapeer, Michigan
  - Karmanos Cancer Institute at McLaren Central Michigan, Morey Cancer Center, Mount Pleasant, Michigan